CLINICAL TRIAL: NCT03820713
Title: Prospective, Randomized, Double Blinded, Parallel, Controlled, Two-arm, Two-center Evaluation of the Feasibility, Safety, Initial Efficacy and Clinical Usability of FuseX Anti-Adhesion System
Brief Title: Evaluation of the Feasibility, Safety, Initial Efficacy and Clinical Usability of FuseX Anti-Adhesion System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eio Biomedical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AOS-CL1000-02; CL-PL-057-01 (Other: EIO Biomedical Ltd.)
Record Dates: First submitted 2018-08-12; First posted 2019-01-29 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Reduction of Postoperative Adhesions
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double blinded, parallel, controlled, two-arm, two-center
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational arm (Experimental): Treatment group receives a concentrate of coagulation factors. The device concentrates coagulation factors from donor plasma; the concentrate is applied to the surgical site intended to reduce the incidence, extent and severity of postoperative adhesions.
  Interventions: Procedure: Concentrate of plasma coagulation factors
- Control arm (Placebo Comparator): Control group receives an identical syringe and applicator generated by processing normal saline 0.9% instead of plasma.
  Interventions: Procedure: 0.9% saline

INTERVENTIONS:
Procedure: Concentrate of plasma coagulation factors — The plasma concentrate of coagulation factors is applied to the surgical site.
  Arms: Investigational arm
Procedure: 0.9% saline — Control group receives an identical syringe and applicator generated by processing normal saline 0.9% instead of plasma.
  Arms: Control arm

SUMMARY:
Evaluation of the feasibility, safety, initial efficacy and usability of FuseX Anti-Adhesion system toward further studies that will be powered to proved its safety and efficacy. In addition, this initial study will serve to yield blood bank and surgeon feedback towards improving the system.

ELIGIBILITY:
Inclusion criteria

PREOPERATIVE INCLUSION

Preoperatively the patient must:

1. Understand and be able to follow the requirements of the protocol including signing and dating an Ethics Committee approved Informed Consent prior to undergoing any protocol related procedures
2. Patients undergoing any of the above procedures
3. Male or female subjects > 18 years of age
4. Subjects for whom a second abdominal surgery is planned within less than 12 months of the first surgical procedure
5. BMI<40

INTRAOPERATIVE INCLUSION

During surgery the patient must require having one of the following surgeries performed on their person:

1. Planned or emergency colonic resection surgery with temporary stoma creation due to colonic perforation, acute diverticulitis or colonic obstruction.
2. Surgery for low rectal cancer - low anterior resection. This surgery includes resection of lower part of rectum, colo-anal anastomosis and protective ileostomy creation. Usually patient undergo second stage procedure closure of ileostomy in 1-3 months.
3. Total proctocolectomy and a pelvic pouch with diverting ileostomy in cases of surgery for Ulcerative colitis. In this kind of surgery there is the intention to close the temporary ileostomy in 1-3 months.
4. Creation of stoma due to infectious process or trauma in the peritoneum (such as Fournier gangrene, laceration of rectum, etc.)

Exclusion Criteria

PREOPERATIVE EXCLUSION

Preoperatively a patient must not:

1. be unable to give their own written informed consent,
2. be currently enrolled in another clinical study with drug or device related to adhesions or has participated in such a study within the last 30 days,
3. have received or is expected to receive any other investigational product or technique belonging to the group of hemostats, adhesion reduction devices or other products, meshes, or other types of implants in the abdominal cavity within 30 days prior to or during enrolment,
4. subjects who have received or will receive (approximately within the next eight months) abdominal/pelvic irradiation for reasons other than rectal carcinoma.
5. BMI≥40
6. Subjects who have received selective factor Xa inhibitors and/or direct thrombin inhibitors within 24 hours prior to surgery.
7. Patients taking immune system suppressants deemed by the surgeon to interfere with wound healing, Patients taking daily doses of corticosteroids exceeding 20mg within the prior 30 days are to be excluded. Patients requiring perioperative corticosteroid supplementation are not to be excluded.
8. Patients with a known history of severe multiple drug allergies
9. Patients who have a life expectancy of less than 6 months because of a medical condition or disease state
10. Any patient with a medical condition or other serious condition which will interfere with compliance and/or ability to complete this study protocol or who in the opinion of the investigator would not be a good candidate for enrollment

INTRAOPERATIVE EXCLUSION

1. Patients for whom it is known, prior to the initial procedure, that loop ileostomy or colostomy closure is not feasible for any reason
2. Patients with peritoneal carcinomatosis
3. Patients with endometriosis
4. Use of hernia mesh in the first surgery.
5. Subjects treated with hemostatic agents in which the sealant remains in the patient's body (e.g. Fibrin sealant).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse event incidence | Within 30 days from the first surgery
  Incidence of adverse events related to treatment requiring any invasive procedure in the test group (who used blood plasma concentrate prepared using FuseX Anti-Adhesion System) compared to control group (who used normal saline processed by the same FuseX Anti-Adhesion System).
Overall adverse event incidence | Until the second surgery but not longer than 7 months
  Overall adverse event incidence will be evaluated by the presence and severity of adverse events and serious adverse events in the test group (who used blood plasma concentrate prepared using FuseX Anti-Adhesion System) vs. control group (who used normal saline processed by the same FuseX Anti-Adhesion System).
Severity of new formed adhesions in the target region | Through study completion, an average of 1 year
  Severity of new formed adhesions having its source in the target region will be assessed by a blinded surgeon during the second surgery by grading the adhesion severity for each region on a scale from 0 (no adhesions) to 3 (strong vascularized adhesions that require sharp dissection and cannot be separated without tissue damage). The peritoneal cavity will be divided into 9 separate scoring regions. A peritoneal adhesion index (PAI) (sum of scores for all the regions) will be calculated per each patient.
Usability as assessed by Surgeon questionnaire | Through study completion, an average of 1 year
  a. Ease of application will be scored on a 5-point Likert scale (1 = very hard to 5 = very easy). b. Percentage of coverage the entire defined surgical field. c. mL of the materials used
Usability as assessed by Operator questionnaire | Through study completion, an average of 1 year
  a. Ease of device use will be scored on a 5-point Likert scale (1 = very hard to 5 = very easy). b. Device operation time

SECONDARY OUTCOMES:
Incidence of general surgical complications; incidence of minor adverse events | Until the second surgery but not longer than 7 months
  Incidence of general surgical complications including but not limited to:
  * Septic shock, cardiovascular events, respiratory tract infections and pulmonary atelectasis, urinary tract infections, thromboembolic events
  * Superficial Surgical Site Infections (SSI) - soft tissue infection, cellulitis, incisional abscess, wound dehiscence
  * Deep SSI - abdominal abscess, pelvic abscess, peritonitis. Incidence of minor adverse events such as nausea, vomiting, abdominal pain, ileus, allergic reactions
Usability of the device Instructions for Use (questionnaire) | Through study completion, an average of 1 year
  Usability of the device user manual will be scored on a 5-point Likert scale (1 = very hard to 5 = very easy).

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Miller, MD, Principal Investigator — EIO Biomedical Ltd., Medical Adviser
Locations (2):
- Lithuania (2):
  - Kaunas Clinical Hospital, Kaunas
  - Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Kaunas